CLINICAL TRIAL: NCT05824416
Title: "Evaluation Of ALBA® Device for Upper Extremity Motor Function In Adults (18-80 Years Old) With Hemiparesis Secondary To Acquired Brain Injury In Subacute And Chronic Phases"
Brief Title: "Evaluation Of ALBA® Device for Upper Extremity Motor Function In Adults With Subacute And Chronic Acquired Brain Injury"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: uMov (Industry)
Collaborators: Clínica los Coihues (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSMOriente030522
Record Dates: First submitted 2023-04-05; First posted 2023-04-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Stroke
Keywords: Stroke; Acquired Brain Injury; Adults
MeSH Terms: conditions — Stroke; Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALBA (Experimental): 25 minutes of therapy with ALBA and 20 minutes with conventional therapy per session for 5 days a week during 4 weeks.
  Interventions: Device: Experimental: ALBA
- Conventional Therapy (Active Comparator): 45 minutes conventional therapy per session for 5 days a week during 4 weeks.
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Device: Experimental: ALBA — Device: Improve Upper Limb Mobility
  The patients will undergo treatment with the conventional therapy, consisting of four types of exercises, including supine and seated exercises, bimanual seated activity, and bipedal exercise. In addition to training with the ALBA® device, Shoulder flexion, abduction, and external rotation, elbow flexion and extension.
  Arms: ALBA
Behavioral: Conventional Therapy — The conventionl therapy will receive conventional treatment, consisting of four types of exercises, including supine and seated exercises, bimanual seated activity, and bipedal exercise
  Arms: Conventional Therapy

SUMMARY:
As part of the rehabilitation techniques, robotic equipment has been introduced for the rehabilitation of the upper extremity with promising results. In this context, the ALBA® devise for the training of the upper extremity is used in this project. This randomized controlled trial will compare a control group (n=16) with an experimental group (n=16) of adults with hemiparesis secondary to an acquired brain lesion. A convenience sample of inpatient will be selected from Los Coihues clinic after concealing the inclusion and exclusion criteria. All participants will perform 45 minutes of training, 5 days a week, for 4 weeks, 20 sessions total. The control group will receive 100% conventional treatment while the experimental group will receive 20 minutes of conventional treatment associated with 25 minutes of ALBA® training. Assessments will be taken before training (t1), at 4 weeks (t2), and at 3 months (t3).

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of occupational therapy for patients with upper limb disabilities, specifically utilizing the ALBA® device for training. Robotic equipment has been introduced as part of rehabilitation techniques for the upper extremity with promising results, and the ALBA® device is being used in this project to assess its effectiveness. A randomized controlled trial will be conducted, comparing a control group receiving conventional treatment and an experimental group receiving a combination of conventional treatment and ALBA® training. Participants will be adults with hemiparesis secondary to an acquired brain lesion, selected from a convenience sample of inpatients at Los Coihues clinic after concealing the inclusion and exclusion criteria.

All participants will perform 45 minutes of training, 5 days a week, for 4 weeks, totaling 20 sessions. The control group will receive 45 minutes of conventional treatment, consisting of four types of exercises, including supine and seated exercises, bimanual seated activity, and bipedal exercise. The experimental group will receive 20 minutes of conventional treatment associated with 25 minutes of supervised ALBA® training. The ALBA® training will involve customizing the device software to the patient's progress and adjusting the angles of inclination for exercises. Each session will feature a virtual assistant guiding patients through a sequence of exercises, including a brief practice period, two series of repetitions of different movements, and a free exercise. Rest periods of 2-3 minutes will be given between each series. Assessments will be taken before training (t1), at 4 weeks (t2), and at 3 months (t3) to evaluate the effectiveness of the two treatment methods. This study design allows for the evaluation of both short and long-term effects. Overall, this study aims to provide evidence for the effectiveness of the ALBA® device for the rehabilitation of upper extremities and contribute to the existing literature on the use of robotic equipment in occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients of Los Coihues clinic Diagnosis of acquired brain injury. Cognitive capacity and language that allows understanding and following the therapist's instructions.

Trunk control. Subacute and chronic stage (up to 2 years post injury). Upper extremity paresis able to perform movements with eliminated gravity (modified MRC 2).

Exclusion Criteria:

Cardiovascular instability Visual or acoustic limitations. Severe hypertonia (≥3 Ashworth Scale). Upper extremity with passive joint limitation and/or traumatic injury. Neuropsychological alteration (global aphasia, severe attentional deficit, spatial perception alteration).

Moderate to severe cognitive-behavioral alterations that do not allow the understanding of instructions.

Severe alterations of consciousness. Deficit in cephalic control. Severe deficit in sedentary balance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-07-11 (Estimated)

PRIMARY OUTCOMES:
Changes on the Fugl-Meyer test | Baseline (t1) and 30 days after (t2)
  The Fugl-Meyer Test is a widely used clinical assessment tool for measuring motor recovery in patients with brain damage, especially after a stroke.
  The test consists of a series of motor activities designed to assess the patient's ability to perform specific movements, such as extending the arm, opening and closing the hand, and standing up from a chair. The movements are scored on a scale of 0 to 2, where 0 means the patient cannot perform the movement and 2 means the patient can perform the movement fully.

SECONDARY OUTCOMES:
ACER-R | Baseline (t1)
  The ACER-R test can be used in the evaluation of individuals who have suffered cognitive damage, such as a stroke or traumatic brain injury. In this case, the test is used to measure cognitive function and determine the degree of cognitive impairment that has occurred.
  In terms of measurement units, the ACER-R uses a standardized scoring system based on the individual's age and the average population score. Scores are expressed in terms of raw scores, standard scores, and percentiles. These scores are used to compare the individual's cognitive capacity with that of the general population and to evaluate the degree of cognitive impairment that has occurred. The minimum possible score is 0 and the maximum is 143.
MRC | Baseline (t1)
  The MRC (Medical Research Council) test is an assessment tool used to measure muscle strength in different muscle groups of the body. It involves the evaluator applying an opposing force to the muscle being evaluated while the individual performs a maximum contraction for several seconds. The strength is measured on a scale of 0 to 5, where 0 indicates a complete absence of muscle contraction and 5 indicates a complete normal contraction.
Ashworth | Baseline (t1)
  The Ashworth test is an assessment tool used to measure muscle tone in people with neurological diseases such as spasticity. It involves evaluating the resistance offered by a muscle to passive movement, i.e. when the evaluator moves the patient's limb in a specific direction without the patient actively participating.
  During the test, the evaluator moves the patient's limb and evaluates the degree of resistance or muscle rigidity on a scale of 0 to 4, where 0 indicates the absence of resistance and 4 indicates severe muscle rigidity. The Ashworth test is used to assess the degree of spasticity in people with brain injuries, cerebral palsy, and other neurological diseases, and can be useful in guiding treatment and rehabilitation.
FIM | Baseline (t1) and 30 days after (t2)
  The FIM (Functional Independence Measure) test is an evaluation tool used to measure functional independence in basic activities of daily living in individuals with physical, neurological, or cognitive disabilities.
  The test consists of an evaluation of 18 items covering six areas of skills: self-care, sphincter control, transfers, locomotion, communication, and cognition. Each item is scored from 1 to 7, where 1 indicates total dependence and 7 indicates total independence.
  The total score is used to determine the individual's level of functional dependence and evaluate the effectiveness of interventions and rehabilitation programs.
Test SF-36 | Baseline (t1), 30 days after (t2) and at follow up (90 days)
  The SF-36 (Short Form-36) is a health survey questionnaire that measures the individual's overall health and quality of life. It consists of 36 questions that assess eight different health domains, including physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. The test is widely used in clinical and research settings to evaluate the impact of health interventions and to compare health outcomes between different populations.
  The SF-36 questionnaire uses a scoring system that ranges from 0 to 100 for each of the eight health domains. A score of 100 indicates the highest level of health or quality of life, while a score of 0 indicates the lowest. Therefore, the total possible score is 800 (100 x 8 domains).
System Usability Scale | Post intervention (30 days)
  The System Usability Scale (SUS) is a questionnaire used to evaluate the usability and user-friendliness of a wide range of technological products, including software, websites, and hardware. The SUS consists of ten questions that assess the user's perception of various aspects of the product's usability, such as its ease of use, efficiency, and learnability. Each question is answered on a five-point scale, ranging from "strongly disagree" to "strongly agree." The SUS score ranges from 0 to 100, with a higher score indicating greater usability and user satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Los Coihues, Santiago, Av. Laguna Sur 6561 Estación Central, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared only in a research framework (e.g., for publication) and on condition of clear acknowledgment of the source by citing the authors. Thus, data will be available upon reasonable request by contacting the corresponding author. The "recipient" must sign a data sharing agreement (DSA) specifying possible (re)uses and the purpose of it.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available starting 6 months after publication

REFERENCES:
- [Derived] Salazar-Cifuentes P, Contreras T, Hernandez E, Leiva-Abarca E, Castro-Flores P, San Juan D, Araneda R, Ebner-Karestinos D. Evaluation of ALBA device for upper extremity motor function in adults with subacute and chronic acquired brain injury: a randomised controlled trial protocol in a tertiary clinic of the metropolitan region of Chile. BMJ Open. 2023 Nov 22;13(11):e076774. doi: 10.1136/bmjopen-2023-076774. PMID 37993168